CLINICAL TRIAL: NCT04275960
Title: An Open-label, Non-randomized, Phase I Study to Evaluate the Pharmacokinetics of Selitrectinib (BAY 2731954) and Food Effects in Healthy Adult Male Participants
Brief Title: Study in Healthy Adult Male Participants to Gather Information How the Human Body Absorbs, Distributes and Excretes the Study Drug Selitrectinib Including the Effect of the Interaction of Food With the Study Drug on the Human Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 21122; 2019-003870-23 (EudraCT Number)
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Solid Tumors Harboring NTRK Fusion
Keywords: Healthy volunteers; Pharmacokinetics; Food-Drug Interactions; Advanced or metastatic solid tumors; Neurotrophic tyrosine receptor kinase (NTRK) gene fusion; Tyrosine receptor kinase (TRK); TRK inhibitor; Drug formulation; Liquid suspension
MeSH Terms: interventions — selitrectinib; Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm_25 + 75 mg (Fasted) (Experimental): Healthy male participants receive a single dose of 25 mg selitrectinib (Period 1) and 75 mg selitrectinib (Period 2) in fasted state.
  Interventions: Drug: Selitrectinib (BAY2731954)
- Arm_50 + 50 mg (Fasted/Fed) (Experimental): Healthy male participants receive a single dose of 50 mg selitrectinib in fasted state (Period 1) and 50 mg selitrectinib in fed state (Period 2).
  Interventions: Drug: Selitrectinib (BAY2731954)
- Arm_100 + 150 mg (Fasted) (Experimental): Healthy male participants receive a single dose of 100 mg selitrectinib (Period 1) and 150 mg selitrectinib (Period 2) in fasted state.
  Interventions: Drug: Selitrectinib (BAY2731954)

INTERVENTIONS:
Drug: Selitrectinib (BAY2731954) — Selitrectinib is administered orally as liquid suspension (20 mg/mL) on Day 1 of each period. Each period lasts 4 days, both periods of each arm are separated by at least 3 days.
  Other Names: Tyrosine receptor kinase (TRK) inhibitor

SUMMARY:
The researchers in this study want to gather information in healthy adult male participants about how the human body absorbs, distributes and excretes the drug selitrectinib including the effect of the interaction of food with the study drug on the human body. Selitrectinib is a new drug under development for the treatment of patients with solid tumor caused by a genetic abnormality known as an NTRK gene fusion which cannot be cured by currently available treatment options or has spread to other parts of the body. The drug blocks the action of the NTRK gene fusion and prevents the activation of certain proteins (TRK fusion proteins), which can cause cancer cells to multiply and form a tumor. Researchers also want to find out if the participants have any medical problems during this study.

Participants in this study will receive the study drug twice with at least 6 days in between. The study drug will be taken orally as a liquid before or after meal. Observation will last for up to 8 weeks, and blood samples will be taken from the participants to measure the blood levels of the study drug.

DETAILED DESCRIPTION:
The primary objectives of this study are to investigate the pharmacokinetics and the effect of food on the pharmacokinetics of selitrectinib after a single dose of the drug.

Secondary objective is to assess the safety of selitrectinib after a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by the investigator or medically qualified designee based on medical evaluation including medical history, laboratory tests, physical, cardiac and neurologic examination
* Body mass index (BMI): ≥18.5 and ≤ 29.9 kg/m2, with body weight ≥50 kg
* Use of adequate contraception until 3 months after last study intervention

Exclusion Criteria:

* Existing relevant diseases of vital organs (e.g. liver diseases, heart diseases), central nervous system (e.g. seizures) or other organs (e.g. diabetes mellitus).
* Medical history of risk factors for Torsades de pointes (e.g. family history of Long QT Syndrome) or other arrhythmias
* Known severe allergies, allergies requiring therapy with corticosteroids, non-allergic drug reactions, or (multiple) drug allergies (excluding untreated asymptomatic seasonal allergies such as non-severe hay fever during the time of study conduct).
* Regular use of medicines
* Regular alcohol consumption
* Smoking more than 5 cigarettes daily
* History of COVID-19 or current SARS-CoV-2 infection

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of selitrectinib in plasma in fasted state (Cmax_fasted) | Up to 3 days
Area under the concentration-time curve of selitrectinib in plasma from time 0 to 24 hours in fasted state (AUC(0-24)_fasted) | Up to 1 day
Area under the concentration-time curve of selitrectinib in plasma from time 0 to infinity in fasted state (AUC_fasted) | Up to 3 days
Maximum concentration of selitrectinib in plasma in fed state (Cmax_fed) | Up to 3 days
Area under the concentration-time curve of selitrectinib in plasma from time 0 to 24 hours in fed state (AUC(0-24)_fed) | Up to 1 days
Area under the concentration-time curve of selitrectinib in plasma from time 0 to infinity in fed state (AUC_fed) | Up to 3 days

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 23 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.